CLINICAL TRIAL: NCT01729689
Title: Intervention Development for Anxiety in Metastatic NSCLC Patients and Their Caregivers
Brief Title: Cognitive Behavioral Therapy in Treating Anxiety in Patients With Stage IV Non-Small Cell Lung Cancer and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ellen Hendriksen, Instructor, Psychiatry & Behavioral Science - Behavioral Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LUN0053; NCI-2012-02096 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25339 (Other: Stanford IRB)
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Anxiety Disorder; Recurrent Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Anxiety Disorders; Carcinoma, Non-Small-Cell Lung | interventions — Counseling

ARMS (1):
- Supportive care (cognitive behavioral therapy) (Experimental): Participants undergo cognitive behavioral therapy over 1 hour once weekly for a total of 6 sessions. Sessions are tailored to patient and caregiver cognitions and approach and avoidance behaviors.
  Interventions: Other: counseling intervention; Other: questionnaire administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Other: counseling intervention — Undergo cognitive behavioral therapy
  Other Names: counseling and communications studies
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This pilot clinical trial studies cognitive behavioral therapy in treating anxiety in patients with stage IV non-small cell lung cancer and their caregivers. Cognitive behavioral therapy may reduce anxiety and improve the well-being and quality of life of patients who have stage IV non-small cell lung cancer and their caregivers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify, through both quantitative and qualitative methods, clinical correlates of anxiety and points of intervention to reduce anxiety in patients with late-stage lung cancer and their primary caregivers.

II. To apply these findings to develop a brief dyadic intervention based on Cognitive Behavioral Therapy (CBT) to reduce anxiety in late-stage lung cancer patients and their primary caregivers.

III. To evaluate the feasibility and acceptability of the pilot intervention through number of completed visits and assessment pre- and post- intervention.

OUTLINE:

Participants undergo cognitive behavioral therapy over 1 hour once weekly for a total of 6 sessions. Sessions are tailored to patient and caregiver cognitions and approach and avoidance behaviors.

After completion of study treatment, participants are followed up at 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage IV non-small cell lung cancer
* At least 6 weeks post-diagnosis
* Current symptoms of anxiety (e.g., Hamilton Rating Scale for Anxiety [HAM-A] >=14)
* Ability to understand and the willingness to sign a written informed consent document
* CAREGIVER: Identified by patient as primary caregiver
* CAREGIVER: At least 14 hours/week spent caring for patient
* CAREGIVER: Current symptoms of anxiety (e.g., HAM-A >= 14)
* CAREGIVER: Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* PATIENTS AND CAREGIVERS:
* Active, unstable, untreated serious mental illness
* Other cognitive inability to complete informed consent process or study procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Feasibility, defined as 75% of participants complete at least 5 sessions, 75% of participants complete pre- and post-intervention assessment battery | Up to 7 weeks
Acceptability, based on qualitative analysis of exit interviews | Up to 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Hendriksen, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States